CLINICAL TRIAL: NCT05810701
Title: FRAGINOC Study: The Impact of FRAilty Screening and Geriatric Assessment and Intervention in Older Patients With Epithelial Ovarian Cancer
Brief Title: FRAGINOC Study: Screening and Geriatric Assessment and Intervention in Older Patients With Epithelial Ovarian Cancer
Acronym: FRAGINOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Herlev Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Tine Henrichsen Schnack, MD, PhD, Associate Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OUHAgeCareOvarian
Record Dates: First submitted 2021-08-25; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer; Frailty
MeSH Terms: conditions — Ovarian Neoplasms; Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: Rancomized clinical trial Combined observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NACT and CGA+ physical training intervention (Active Comparator): Elderly (≥70 years) ovarian cancer patients referred for Neo-adjuvant treatment randomized to comprehensive geriatric assessment and individualised physical training.
  Interventions: Other: Comprehensive geriatric assessment and individualised physical training
- NACT no intervention (No Intervention): Elderly (≥70 years) ovarian cancer patients referred for Neo-adjuvant treatment randomized to standard of care

INTERVENTIONS:
Other: Comprehensive geriatric assessment and individualised physical training — Comprehensive geriatric assessment and relevant intervention (including medical and pharmacological optimisation, nutritional, social and psychological intervention, among others), and individualised physical training
  Arms: NACT and CGA+ physical training intervention

SUMMARY:
Ovarian cancer (OC) is the fifth most common cause of cancer death. More than 40% are older than 70 years. The standard treatment is radical surgery combined with chemotherapy. More than 40% of the Danish patients will never undergo surgery. Frail and immunodeficient older patients are at higher risk of complications, and immunomodulating treatment as chemotherapy results in different outcomes in comparable patients. No accurate validated screening tool to identify frail and immunodeficient OC women exists. Optimization through comprehensive geriatric assessment (CGA) and physical training before and during treatment may improve outcomes and decrease associated risks.

Aim: Primary endpoints will be to determine whether a CGA and physical training vs standard of care can increase the proportion of patients later on referred to interval debulking surgery, and examine the performance of validated screening tests in predicting impairments in CGA. Other endpoints will be to evaluate if intervention can improve completion of chemotherapy, to examine the association between frailty screening scores and selected biomarkers with treatment outcomes, including complications and quality of life, and ultimately to develop an improved frailty screening tool based on known screening tools, functional tests and biomarkers identifying patients who will benefit from CGA.

Method: This is a nationwide, randomized intervention study. Patients ≥70 years diagnosed with primary OC at the Gynecological departments of Rigshospitalet, Odense and Roskilde University Hospitals will be included. In an interdisciplinary collaboration between medical specialists in oncology, gynecology and geriatrics, included patients will be screened for frailty using validated screening tools and functional tests. Specific biomarkers and immunologic profile will be assessed in all patients. Patients selected for neoadjuvant chemotherapy will be randomized to receive CGA or standard of care. Patients selected for primary debulking surgery or palliation will be followed in an observational cohort.

Perspective: The development of a validated screening tool for frailty assessment and immunological status will help us identify frail patients who may need optimization before treatment, resulting in more patients getting optimal treatment (either surgery or chemotherapy), prevent post-treatment complications and avoid palliative patients from undergoing a redundant complex treatment.

DETAILED DESCRIPTION:
Introduction

Several studies have shown that a high percentage of patients with epithelial ovarian cancer (EOC) are undertreated due to their age, even in the absence of comorbidity. On the other hand, there seems to exist a group of frail patients unfit for extensive treatment that are over-treated. Therefore, it is of great interest to identify the group of older patients with EOC, who are frail and would benefit of a comprehensive geriatric assessment and optimisation, including individualised physical training. Unfortunately, no specific screening tool can be recommended or discouraged, and none of these tests are validated in patients with EOC.

Immunodeficiency and biomarkers regarding nutritional status, strength, and general health are not part of the standard evaluation, although several studies have shown a correlation between these factors and the functional independence of older patients, comorbidity, postoperative complications, tolerance to chemotherapy and quality of life.

In oncologic geriatrics a Comprehensive Geriatric Assessment (CGA - an examination performed by an interdisciplinary geriatric team) can be performed before start of treatment. Unfortunately, a complete CGA is both time and resource consuming, and the impact of interventions in older patients with EOC has never been examined.

Hypothesis and purpose

Our hypothesis is that frail patients with advanced ovarian cancer can benefit from a geriatric assessment and optimization, including physical training, increasing their chances of referral to surgery and to get full oncological treatment. The investigators believe that it is possible to develop a frailty screening tool with highly improved accuracy by combining known frailty screening tests, functional tests, and relevant biomarkers, which can help us select those patients who will benefit from a geriatric assessment and intervention.

The clinical study is parceled out in two working projects, WP1 and WP2, which are anchored at the departments of gynecology, geriatric medicine, and oncology at several centers in Denmark.

- WP1: Geriatric assessment and intervention and its impact on treatment outcomes examined in a cohort of older patients with EOC referred to NACT Primary endpoint: To determine whether a CGA and tailored intervention vs. standard of care can increase the proportion of patients referred to IDS.

Secondary endpoints are a)to evaluate whether a CGA and tailored intervention can improve completion of chemotherapy, b) to investigate if CGA and a tailored intervention with physical training vs. standard of care improves treatment outcome and quality of life.

- WP2: Impact of biomarkers, functional tests and immunological profile in assessing frailty and as predictors of adverse treatment outcomes in a national cohort of older EOC patients.

Primary endpoint: to examine the performance of three validated frailty screening tests (G8, mG8, and Clinical Frailty Index (CFI)) in EOC patients in predicting impairments in CGA.

Secondary endpoints are a)to examine whether adding functional tests, biomarkers, and the immunological profile can improve the accuracy of the frailty screening tests b) to examine whether the screening tool is predictive of patients achieving radical surgery and completing oncological treatment, as well as predict adverse treatment outcomes

Method description

The FRAGINOC project is a multicenter study, where WP1 is a clinical randomized trial of screening and intervention in older patients (≥70 years) with a diagnose of advanced EOC (FIGO stage III-IV). WP2 is a prospective observational study, where patients from WP1 will be asked to participate. Furthermore, older patients (≥70 years) referred to PDS or palliation will also be included. Patients will be evaluated at MDT conference, where they will be referred to either PDS and chemotherapy or NACT or palliation. Those referred to NACT will be re-evaluated at a second MDT conference after three cycles of chemotherapy to decide whether they can be referred to IDS.

Screening

All included patients will be screened for frailty after the MDT conference using a combination of the following tools:

* Questionnaires (Geriatric-8, modified Geriatric-8 and clinical frailty scale).
* Functional tests (hand grip test, 30 second chair test and 6 minutes walk test)
* Blood samples, which have all been validated previously although in other cancer types.

These tests will be repeated after the second MDT conference (after 3rd cycle of chemotherapy or before interval surgery)

Randomization and Intervention After the initial frailty screening, patients eligible for primary chemotherapy will be randomized 1:1 to CGA and tailored intervention or standard of care.

The intervention group will be evaluated by a geriatric specialist team examining different domains of their health status with the help of different validated questionnaires and tests, and tailored interventions will be made according to identified needs in the assessed health domains following the geriatric evaluation.

The intervention will specifically include a tailored-made physiotherapy training program of around 9-12 weeks duration, available in both physical and virtual versions. The program consists on supervised resistance training two days a week, either at hospital appointments or virtually from the patients' own home. Those patients who are not able to make the virtual training will be followed up by phone twice a week by the physiotherapist. Additionally, the training will be supported by a progressive walking program measured with a Garmin Vivofit 4 activity tracker. Patients will be thoroughly assessed by a physiotherapist during the training process. Nutritional supplements and advice on sufficient nutrition will be provided according to current clinical guidelines.

Patient-reported outcomes Measures (PROMs) All patients will be asked to complete the European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire - Ovarian Cancer Module (EORTC QLQ C-30, QLQ-OV28) and the supplemental Elderly Cancer Patients Module questionnaire (ELD-14), as well as European Quality of Life- 5 dimensions- 5 levels questionnaire (EQ-5D-5L for cost-utility analysis, at inclusion, after three cycles of chemotherapy, and at the end of treatment.

When assessing the quality of recovery, the QoR-15 questionnaire will be used and evaluated before surgery and 72 hours after PDS or IDS.

Statistical plan/recruitment consideration According to the literature and clinical experience, increasing the number of patients who receive surgery from the present 57 % to 77 % is clinically relevant and possible. To detect a difference of 20 % and obtain a type I error rate of 5% and a power of 80%, a sample size of 86 patients per study arm will be needed. To account for an expected dropout rate of ~20%, it was decided to increase this number to a group size of 100. Thus, a total of 206 patients referred to NACT will be included in the study (WP1 only). Patients referred to PDS will be followed in an observational design. For the last three years, 130 patients fulfilling the inclusion criteria have been treated at RH, OUH, HUH, and SUH each year. Thus, inclusion is expected to run over 2-3 years.

Data will be collected prospectively (demographic, clinical, pathologic, and results from frailty screening, functional tests, blood tests, and intervention effects), and recorded in predesigned RedCap. PRO will be completed by the patients either electronically and registered directly in RedCap, by phone calls or delivered in hand to the Ph.D. student or research nurses. Life-long follow-up data on overall survival will be obtained from the Danish Hospital Registry through linkage with a personal identification number.

Logistic regression will be used to evaluate change over time in ordinal categorical values. Independent T-tests will be used to evaluate in-group and between-groups differences. Kaplan-Meier method and Cox regression analyses will be used to analyze Progression Free Survival.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ovarian cancer
* Capable of understanding written and oral danish

Exclusion Criteria:

* Other active cancers in the preceding 5 years
* Severe psychiatric disease

Patients referred to primary debulking surgery will be followed in a observational design

Ages: 70 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Women as only women are diagnosed with ovarian cancer
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Interval Debulking Surgery | Up to 8 months
  Proportion of patients referred to interval debulking surgery
Frailty screening questionnaires | Up to 8 months
  Specificity and positive and negative predictive values of Geriatric-8, modified Geriatric-8 and Clinical Frailty Scale, in predicting impairments in Comprehensive Geriatric assessment

SECONDARY OUTCOMES:
Completion of chemotherapy treatment | Up to 8 months
  Proportion of patients who complete oncological treatment (≥90% of the intended treatment)
Effect of training: Physical capacity and endurance | Up to 8 months
  Median of score result in meters of Six-Minute-Walk-Test
Effect of training: Physical function and strength | Up to 8 months
  Median of score result of 30 sec Sit-to-Stand Test in number (lower body) and of Hand Grip Strength test in Kg (upper body)
Effect of physical training: Physical function in relation to basic mobility | Up to 8 months
  Median of Timed Up and Go test in seconds
Effect of physical training: Physical function in relation to balance | Up to 8 months
  Median of Guralnik test: score in seconds
Effect of physical training: Clinical reported measurements | Up to 8 months
  Median of Performance status (number 0-4), Clinical Frailty Scale (1-9), G8 ( 0-17) and modified G8 (0-35)
Effect of physical training: Self-reported measurements | Up to 8 months
  Median of ELFI (0-100), Physical fitness (1-5) and FES-1 short (7-28)
Patient-reported outcomes measures (PROMs) | Up to 8 months
  Median of score of quality of life and recovery questionnaires
Frailty screening combined tool | Up to 8 months
  Specificity and positive and negative predictive values of a combination of Handgrip strength test, 30 second-chair stand test and 6 minutes walk tests, as well as serum concentrations of inflammatory biomarkers added to screening questionnaires (G8, mG8 and CFS), in predicting impairments in Comprehensive Geriatric assessment
Postoperative complications | Up to 8 months
  Median of score of Clavien-Dindo of complications within 30 days after surgery
Progression Free-Survival | Up to 2 years
  Median of period of time measured in months without recurrence of ovarian cancer

OTHER OUTCOMES:
Comprehensive Geriatric Assessment | Up to 8 months
  Rate of number of intervened domains
Hospital admissions related to chemotherapy | Up to 8 months
  Rate of number and length of hospital admissions during chemotherapy treatment
Physical activity in intervention group-walking | Up to 8 months
  Median of daily distance in meters measured by an activity tracker
Physical activity in intervention group-training | Up to 8 months
  Rate of completion of training intervention
Radicality of Surgery | Up to 8 months
  Rate of optimal debulking vs suboptimal debulking during surgery
Inflammatory biomarkers | Up to 8 months
  Median of serum concentrations of inflammatory biomarkers (CRP, IL-6, YKL-40 and a panel of 92 proteins)
Sarcopenic biomarkers | Up to 8 months
  Median of serum concentrations of GDF-11 and GDF-15

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Odense University Hospital, Odense, Region of South Denmark
  - Vejle Hospital, Vejle, Region of South Denmark
  - Zealand University Hospital, Roskilde, Region Sjælland
  - Copenhagen University Hospital Rigshospitalet, Copenhagen, The Capital Region of Denmark
  - Herlev and Gentofte Hospital, Herlev, The Capital Region of Denmark

IPD SHARING:
Plan to Share IPD: No
We do plan to make data available to other researchers but have not yet decided how